CLINICAL TRIAL: NCT03694366
Title: Integrated Community Based Health Systems Strengthening in Northern Togo: A Stepped-Wedge Randomized Cluster Pragmatic Control Trial
Brief Title: Integrated Community Based Health Systems Strengthening in Northern Togo
Acronym: ICBHSS-Togo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Integrate Health (Other)
Collaborators: Ministère de la Santé et de l'Hygiène Publique, Togo (Unknown); Université de Lomé, Faculté des Sciences de la Santé, Togo (Unknown); Albert Einstein College of Medicine (Other); Montefiore Medical Center (Other); City University of New York, School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: ICBHSS
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Maternal and Child Health; Health Service Utilization
Keywords: Child Mortality; Reproductive, Maternal, Newborn, and Child Health; Community Health Workers; Implementation Research; Health Systems Strengthening
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Five facilities in Bassar District: Estimated population of 34,676 served by five public sector facilities in Bassar District.
  Interventions: Other: ICBHSS model
- Seven facilities in Binah District: Estimated population of 31,027 served by seven public sector facilities in Binah District.
  Interventions: Other: ICBHSS model
- Four facilities in Dankpen District: Estimated total population of 40,165 served by four public sector facilities in Dankpen District.
  Interventions: Other: ICBHSS model
- Five facilities in Kéran District: Estimated total population of 31,866 served by five public sector facilities in Kéran District.
  Interventions: Other: ICBHSS model

INTERVENTIONS:
Other: ICBHSS model — Bundle of evidence-based interventions that include the following 5 components:
  1. Community engagement meetings and feedback;
  2. Elimination of public sector facility user fees for children under five and pregnant women;
  3. Pro-active community based IMCI using trained, equipped, supervised, and salaried Community Health Workers (CHWs) with additional services including linkage to family planning and counseling, HIV testing & referrals;
  4. Clinical mentoring and enhanced supervision by a trained peer coach at public sector facilities;
  5. Basic infrastructure improvements and supply chain management training of pharmacy managers

SUMMARY:
The general objective of this study is to optimize implementation and assess effectiveness of the integrated facility and community-based health systems strengthening (ICBHSS) model in four Northern Togo districts, using the RE-AIM implementation science framework. Specific study aims include: (1) Analyze longitudinal changes regarding maternal and child health outcomes, health service utilization rates, and public sector facility readiness in the ICBHSS model intervention sites catchment areas; (2) Identify barriers to and facilitators of access and quality services related to ICBHSS model; and (3) Assess changes in health care services coverage, effectiveness, and adoption of ICBHSS model. These findings are expected to contribute to continuous quality improvement initiatives, optimize implementation factors, provide generalizable knowledge regarding health service delivery, and accelerate health systems improvements in Togo and more broadly.

DETAILED DESCRIPTION:
Background: Over the past decade the burden of poor maternal and child health outcomes in Togo, particularly in the Northern regions, have remained high despite global progress. The principal causes of under-5 deaths in Togo are diseases with effective and low-cost prevention and or treatment strategies, including malaria (18%), acute lower respiratory infections (15%), and diarrheal diseases (8%).While Togo has an official plan for the integrated management of childhood illness (IMCI), including a permissive policy on integrated community case management (iCCM), challenges in implementation persist with low public sector health service utilization.There are critical gaps in access and quality of community health systems throughout the country and an urgent need to improve health outcomes through expanding access and quality of services.

Intervention: The investigators have adapted an integrated facility and community-based health systems strengthening (ICBHSS) model to improve primary healthcare services in Togo. The ICBHSS model includes a bundle of evidence based interventions including (1) community engagement meetings and feedback; (2) the elimination of facility user fees for children under five and pregnant women; (3) pro-active community based IMCI using Community Health Workers (CHWs) with additional services including linkage to family planning and counseling, HIV testing & referrals; (4) clinical mentoring and enhanced supervision at public sector facilities; and (5) improved supply chain management and facility structures. In 2015, a pilot ICBHSS initiative was launched in partnership with the Ministry of Health (MOH) at four public sector clinics in Northern Togo. Preliminary results from this pilot intervention suggested a meaningful reduction in children under-5 deaths, with a trend in reduction for under-one deaths as well as increased health service utilization at all 4 sites. In collaboration with MOH and technical partners, IH developed a plan to expand the ICBHSS model to 21 distinct health facilities over a four-year period in four additional districts: Bassar, Binah, Dankpen, and Kéran. The planned roll out includes expanding into a new district every 12 months based on budgetary and feasibility considerations. As part of this expansion planned for 2018, Integrate Health (IH) and MOH partners are planning an implementation study to both improve service delivery at expansion sites and inform national scale strategies.

Study: The investigators will conduct a mixed methods assessment, using the RE-AIM framework to evaluate the impact and implementation of the ICBHSS initiative in 4 districts. Consists of three key components: (1) a stepped-wedge randomized cluster pragmatic control trial to obtain annual coverage, effectiveness, and adoption metrics using a population-based household survey, (2) health facility assessments to be completed at the cluster (district) level for each health facility prior to intervention launch and post-intervention, and (3) key informant interviews conducted at 12, 24, 48 months for each cluster. The primary outcome will be under 5 year old mortality rate, with secondary outcomes including under-one mortality rate, maternal mortality rate, as well as maternal and child health service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Female of reproductive age (aged 15-49 years)
* Individuals aged 15-17 years will only be included if they have children and/or are pregnant
* Lives in selected household within study catchment area
* Informed consent is obtained for participants 18-49
* Waiver of parental permission is obtained for 15-17 year-old participants

Exclusion Criteria:

* None

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Females of reproductive age (aged 15-49 years) who reside in a selected household within the study catchment area.
Sampling Method: Probability Sample
Enrollment: 7600 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Under-five year old mortality rate | 48 months
  The under-five mortality rate (expressed as a rate per 1,000 live births) is the probability of a child dying in a specified year between birth and 5 years of age.

SECONDARY OUTCOMES:
Under-one year old mortality rate | 48 months
  The under-one mortality rate (expressed as a rate per 1,000 live births) is the probability of a child dying in a specified year between birth and 1 year of age.
Maternal mortality rate | 48 months
  The maternal mortality rate (expressed as a rate per 100,000 live births) is the probability of a mother dying in a specified year within 42 days of pregnancy termination .
Proportion of children under age five reported to be febrile in the prior two weeks who received an effective antimalarial treatment within 24 hours of symptom onset. | 48 months
  The number of febrile children under-five who received an effective antimalarial treatment within 24 hours of symptom onset out of the total number of children under age five reported to be febrile in the prior two weeks.
Proportion of children under age five reported to have a cough in the prior two weeks who received an effective pneumonia treatment within 24 hours of symptom onset. | 48 months
  The number of children under-five who received an effective pneumonia treatment within 24 hours of symptom onset out of the total number of children under age five reported to have a cough in the prior two weeks.
Proportion of children under age five reported to have diarrhea in the prior two weeks who received an effective treatment for diarrheal disease within 24 hours of symptom onset. | 48 months
  The number of children under-five who received an effective treatment for diarrheal disease within 24 hours of symptom onset out of the total number of children under age five reported to have diarrhea in the prior two weeks.
Maternal facility based birth delivery incidence rate | 48 months
  The proportion of women reported to have delivered in a health facility.
Protocol Adherence by IH community health workers in iCCM and maternal consultations | 48 months
  The average adherence by IH community health workers to evidence based protocols for iCCM and maternal consultations.
Protocol adherence by clinical staff at IH intervention facilities in iCCM and maternal consultations | 48 months
  The average adherence by public sector clinical staff at IH intervention sites to evidence based protocols for iCCM and maternal consultations.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Fiori, Jr., MD, MPH, Principal Investigator — Integrate Health; Albert Einstein School of Medicine; Molly E Lauria, MPH, Study Director — Integrate Health
Locations (1):
- Integrate Health, Kara, Togo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiori K, Schechter J, Dey M, Braganza S, Rhatigan J, Houndenou S, Gbeleou C, Palerbo E, Tchangani E, Lopez A, Bensen E, Hirschhorn LR. Closing the delivery gaps in pediatric HIV care in Togo, West Africa: using the care delivery value chain framework to direct quality improvement. AIDS Care. 2016 Mar;28 Suppl 2(sup2):29-33. doi: 10.1080/09540121.2016.1176678. PMID 27391996
- [Background] McCarthy KJ, Braganza S, Fiori K, Gbeleou C, Kpakpo V, Lopez A, Schechter J, Singham Goodwin A, Jones HE. Identifying inequities in maternal and child health through risk stratification to inform health systems strengthening in Northern Togo. PLoS One. 2017 Mar 16;12(3):e0173445. doi: 10.1371/journal.pone.0173445. eCollection 2017. PMID 28301539
- [Derived] Lauria ME, Fiori KP, Jones HE, Gbeleou S, Kenkou K, Agoro S, Agbere AD, Lue KD, Hirschhorn LR. Assessing the Integrated Community-Based Health Systems Strengthening initiative in northern Togo: a pragmatic effectiveness-implementation study protocol. Implement Sci. 2019 Oct 16;14(1):92. doi: 10.1186/s13012-019-0921-3. PMID 31619250
- See also: Integrate Health — https://integratehealth.org/